CLINICAL TRIAL: NCT00860093
Title: A Multi-Site Placebo-Controlled Randomized Double-Blind Study to Evaluate the Efficacy and Safety of Using MPC-5971 as Adjuvant Therapy in Subjects Undergoing Shock Wave Lithotripsy
Brief Title: Efficacy and Safety of Using MPC-5971 in Subjects Undergoing Shock Wave Lithotripsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Corporate Business Decision
Sponsor: Mission Pharmacal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MPC-5971
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Nephrolithiasis
Keywords: Kidney Calculi; Urolithiasis; Lithotripsy; potassium compounds; magnesium compounds
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi; Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): MPC-5971
  Interventions: Drug: MPC-5971
- 2 (Placebo Comparator): placebo identical in appearance to study drug
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — After SWL treatment subjects will be randomized to receive either MPC-5971 or placebo. Two tablets of MPC-5971 or placebo will be taken orally twice a day (bid). This will give a daily dosage equal to 40 mEq of potassium, 20 mEq of magnesium and 60 mEq of citrate. MPC-5971 or placebo will be taken bid for 90 days beginning immediately after SWL treatment.
  Arms: 2
Drug: MPC-5971 — After SWL treatment subjects will be randomized to receive either MPC-5971 or placebo. Two tablets of MPC-5971 or placebo will be taken orally twice a day (bid). This will give a daily dosage equal to 40 mEq of potassium, 20 mEq of magnesium and 60 mEq of citrate. MPC-5971 or placebo will be taken bid for 90 days beginning immediately after SWL treatment.
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the efficacy of MP-5971 in facilitating stone passage after Shock Wave Lithotripsy treatment.

DETAILED DESCRIPTION:
Shock Wave Lithotripsy (SWL) is widely utilized as a first line therapy in patients with renal calculi. SWL is associated with limited morbidity, however, complications relating to stone fragment passage after treatment can occur, the most serious being ureter obstruction. In addition, the growth and agglomeration of residual fragments after SWL treatment, in approximately 40% of patients, will lead to another stone episode within 12 months. Adjunct therapy with MPC-5971 should reduce the risk of complications of residual stone fragments by facilitating passage, preventing blockage and inhibiting growth and enlargement of residual fragments. This is based on MPC-5971's ability to increase urinary inhibitors against growth and agglomeration of stone fragments and by reducing urinary saturation of calcium oxalate and uric acid. The objective is to see a decrease in fragment complications and a significant increase in the stone free rate at 3 months following SWL treatment in combination with MPC-5971.

ELIGIBILITY:
Inclusion criteria:

* Male or female subject aged > or equal to 18 to < or equal to 70.
* Subject has undergone a computerized tomography (CT) scan within 30 days of the screening visit.
* Subject has been diagnosed with single unilateral renal calculus (target treatment stone).
* Target treatment stone, is presumed to be of calcium composition and/or uric acid composition.
* Target treatment stone is between > or equal to 5 and < or equal to 15 mm in diameter.
* Contra lateral kidney may hold a clinically inconsequential size calculus that does not require concurrent SWL treatment.
* Both kidneys are anatomically normal.
* An appropriate candidate for SWL, determined by treating physician.
* Female subjects with a negative pregnancy test, hysterectomy, tubal ligation or non-child bearing potential (post-menopausal).
* Female subjects of child bearing potential with a negative pregnancy test and taking appropriate birth control for the duration of the study.
* Urine is pyuria negative and nitrite negative on dipstick and/or negative upon microscopic evaluation.
* Subject must voluntarily consent to participate in this study and provide his/her written informed consent prior to start of any study-specific procedures.

Exclusion Criteria:

* Current or past history of cystine stones or infection stones.
* Renal insufficiency, defined as serum creatinine value outside of the normal reference range.
* Currently has or had hyperkalemia within the past six months, defined as serum potassium outside of the normal reference range.
* Currently has or had hypermagnesemia within the past six months, defined as serum magnesium outside of the normal reference range.
* Active urinary tract infection.
* Renal calculi in an anatomically abnormal kidney; horseshoe shape, ureteropelvic junction obstruction or calyceal diverticulum.
* Altered urinary tract anatomy such as a transplant kidney, urinary reconstruction or congenital anomaly.
* Blood coagulopathies and or taking anticoagulants (warfarin, coumarin, heparin).
* Taking salicylate (aspirin), including low dose aspirin for cardio-prophylaxis or other NSAID (OTC) that may increase bleeding time, within the past 7 days.
* History of complications with previous SWL; pyelonephritis, perinephric hematoma.
* Unsuccessful SWL treatments for previous stone within the past six months.
* Currently has or previously had ulcers of the esophagus, stomach and/or small intestines.
* Chronic diarrhea or has a history of diarrhea.
* Bowel disease such as Crohn's disease, Celiac disease, fat malabsorption or Sprue.
* Undergone any bariatric surgery procedures.
* Obese, defined as BMI >30.
* Uncontrolled hypertension defined as subjects taking medication specific for hypertension or subject not on medication with systolic blood pressure above 140 and diastolic above 90.
* Adrenal insufficiency (i.e., Addison's disease), adrenal tumors, and/or subjects on adrenal hormone replacement therapy.
* Taking potassium-sparing diuretics (triamterene, amiloride, spironolactone, Midamor®, Aldactone®, Dyrenium®, Eplerenone®).
* Taking potassium supplements (Rx or OTC) within the past 15 days.
* Taking magnesium supplements (Rx or OTC) within the past 15 days.
* Taken potassium citrate supplements (Rx or OTC) within the past 30 days.
* Subject taking anticholinergic medications at entry (dicyclomine, atropine, scopolamine, oxybutynin, tolerodine, Cogentin®, Sinemet®, Robinal®, Kenadrin®, Artane®, Enablex®, Detrol®, Vesicare®, Sanctura®, Ditropan®, Oxytrol®, Bentyl®, Byclomine®, Dibent®, Di-Spaz®, or Dilomine®). (Subjects may be prescribed anticholinergics as standard of care with use of stents post entry.)
* Subject is has taken gastrointestinal enzyme replacement therapy or proton pump inhibitors within past 30 days (Ultrase®, Creon®, Viokase®, Pancrease® MT, pancrelipase agents, Aciphex®, Nexium®, Prevacid®, Protonix®, Zegerid® Prilosec OTC®, Kapidex®, rabeprazole, esomeprazole, lansoprazole, pantoprazole, omeprazole, dexlansoprazole).
* Women who are pregnant or lactating.
* Subjects with a known hypersensitivity to potassium, magnesium, citrate or any excipients in the drug formulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
stone free rate after SWL treatment | 12 weeks

SECONDARY OUTCOMES:
increase in urine inhibitors | 4 week and 12 week
Reduced need for secondary procedures such as URS to clear obstructive fragments | 12 weeks
reduced stone/fragment area (mm2),percent change from the treatment stone area (mm2) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Idaho Urologic Institute, Meridian, Idaho
  - Columbus Urology Research, Columbus, Ohio
  - Urology Clinics of North Texas, PA, Dallas, Texas

REFERENCES:
- [Background] Koenig K, Padalino P, Alexandrides G, Pak CY. Bioavailability of potassium and magnesium, and citraturic response from potassium-magnesium citrate. J Urol. 1991 Feb;145(2):330-4. doi: 10.1016/s0022-5347(17)38330-1. PMID 1988724
- [Background] Pak CY, Koenig K, Khan R, Haynes S, Padalino P. Physicochemical action of potassium-magnesium citrate in nephrolithiasis. J Bone Miner Res. 1992 Mar;7(3):281-5. doi: 10.1002/jbmr.5650070306. PMID 1585829
- [Background] Ettinger B, Pak CY, Citron JT, Thomas C, Adams-Huet B, Vangessel A. Potassium-magnesium citrate is an effective prophylaxis against recurrent calcium oxalate nephrolithiasis. J Urol. 1997 Dec;158(6):2069-73. doi: 10.1016/s0022-5347(01)68155-2. PMID 9366314
- [Background] Gonzalez GB, Pak CY, Adams-Huet B, Taylor R, Bilhartz LE. Effect of potassium-magnesium citrate on upper gastrointestinal mucosa. Aliment Pharmacol Ther. 1998 Jan;12(1):105-10. doi: 10.1046/j.1365-2036.1998.00280.x. PMID 9692708
- [Background] Ruml LA, Wuermser LA, Poindexter J, Pak CY. The effect of varying molar ratios of potassium-magnesium citrate on thiazide-induced hypokalemia and magnesium loss. J Clin Pharmacol. 1998 Nov;38(11):1035-41. doi: 10.1177/009127009803801108. PMID 9824785
- [Background] Ruml LA, Gonzalez G, Taylor R, Wuermser LA, Pak CY. Effect of varying doses of potassium-magnesium citrate on thiazide-induced hypokalemia and magnesium loss. Am J Ther. 1999 Jan;6(1):45-50. doi: 10.1097/00045391-199901000-00007. PMID 10423646
- [Background] Ruml LA, Pak CY. Effect of potassium magnesium citrate on thiazide-induced hypokalemia and magnesium loss. Am J Kidney Dis. 1999 Jul;34(1):107-13. doi: 10.1016/s0272-6386(99)70115-0. PMID 10401023
- [Background] Wuermser LA, Reilly C, Poindexter JR, Sakhaee K, Pak CY. Potassium-magnesium citrate versus potassium chloride in thiazide-induced hypokalemia. Kidney Int. 2000 Feb;57(2):607-12. doi: 10.1046/j.1523-1755.2000.00881.x. PMID 10652038
- [Background] Jaipakdee S, Prasongwatana V, Premgamone A, Reungjui S, Tosukhowong P, Tungsanga K, Suwantrai S, Noppawinyoowong C, Maskasame S, Sriboonlue P. The effects of potassium and magnesium supplementations on urinary risk factors of renal stone patients. J Med Assoc Thai. 2004 Mar;87(3):255-63. PMID 15117041
- [Background] Tosukhowong P, Tungsanga K, Phongudom S, Sriboonlue P. Effects of potassium-magnesium citrate supplementation on cytosolic ATP citrate lyase and mitochondrial aconitase activity in leukocytes: a window on renal citrate metabolism. Int J Urol. 2005 Feb;12(2):140-4. doi: 10.1111/j.1442-2042.2005.01001.x. PMID 15733107
- [Background] Sriboonlue P, Jaipakdee S, Jirakulsomchok D, Mairiang E, Tosukhowong P, Prasongwatana V, Savok S. Changes in erythrocyte contents of potassium, sodium and magnesium and Na, K-pump activity after the administration of potassium and magnesium salts. J Med Assoc Thai. 2004 Dec;87(12):1506-12. PMID 15822549
- [Background] Odvina CV, Mason RP, Pak CY. Prevention of thiazide-induced hypokalemia without magnesium depletion by potassium-magnesium-citrate. Am J Ther. 2006 Mar-Apr;13(2):101-8. doi: 10.1097/01.mjt.0000149922.16098.c0. PMID 16645424
- [Background] Zerwekh JE, Odvina CV, Wuermser LA, Pak CY. Reduction of renal stone risk by potassium-magnesium citrate during 5 weeks of bed rest. J Urol. 2007 Jun;177(6):2179-84. doi: 10.1016/j.juro.2007.01.156. PMID 17509313